CLINICAL TRIAL: NCT05036044
Title: An Observational Cohort Study of Associations Between Early Neurological Complications（including Stroke）and Carotid-Cerebral Vascular Disease Among Patients After Coronary Artery Bypass Grafting
Brief Title: Stroke and Carotid-Cerebral Vascular Disease After CABG
Acronym: SCCAB
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and Director, Department of Cardiovascular Surgery, Vice President, Ruijin Hospital, Ruijin Hospital
Other Study IDs: KY-2021127
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Bypass
Keywords: Neurological complications; Carotid-cerebral artery disease; CABG; CAD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With moderate or severe carotid-cerebral artery disease: moderate (stenosis 50-69%) or severe (stenosis 70-100%) carotid-cerebral artery disease
- Without moderate or severe carotid-cerebral artery disease: mild (stenosis 30-49%) or no (stenosis 0-29%) carotid-cerebral artery disease

SUMMARY:
Review the data of patients who underwent coronary artery bypass grafting (CABG) at the Department of Cardiovascular Surgery in Ruijin hospital from March 2020 to May 2022, including medical history, head and neck CTA, head CT scan, and early postoperative (within 7 days after surgery) neurological complications (defined as a composite of stroke, delayed awakening and severe delirium) . Case-control and retrospective cohorts were built to explore risk factors of early postoperative neurological complications, And its association with baseline carotid-cerebral vascular disease.

Describe the epidemiological data of early postoperative neurological complications (stroke, delayed awakening, and severe delirium) after CABG surgery (within 7 days after surgery); explore independent risk factors of compound neurological complications, build predictive models; compare the effects of carotid-cerebral artery disease on early postoperative compound neurological complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received CABG at the department of cardiac surgery in our hospital.
2. Surgery that patients received includes both isolated and combined CABG surgery.
3. Includes both cardiopulmonary and non-cardiopulmonary bypass.

Exclusion Criteria:

1. Without complete preoperative examination data, such as carotid-cerebral artery CTA, head CT imaging results and so on.
2. Without complete baseline medical history and 7 day post-surgery record.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients received CABG at the department of cardiac surgery in Ruijin hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
the incidence of 7-day neurological complications | within 7 days post-CABG
  a composite of stroke, delayed awakening, severe delirium
the incidence of 7-day stroke | within 7 days post-CABG
  including cerebral infarction, cerebral hemorrhage, and hypoxic-ischemic encephalopathy
the incidence of delayed awakening | within 48 hours post-CABG
  post-surgery patient does not wake up at 48 hours after withdrawing sedative
the incidence of severe delirium | within 7 days post-CABG
  ICU CAM-II score≥2 points

SECONDARY OUTCOMES:
the incidence of All-cause death | 7 days, 30 days and 1 year post-CABG
  Death from any cause
the incidence of CV-death | 7 days, 30 days and 1 year post-CABG
  Including death resulting from an acute myocardial infarction , sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular procedures, death due to cardiovascular hemorrhage, and death due to other cardiovascular causes
the incidence of myocardial infraction | 7 days, 30 days and 1 year post-CABG
  According to the 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials, including CABG-related MI, non CABG-related MI, silent MI and unknown type.
the incidence of repeat revascularization | 7 days, 30 days and 1 year post-CABG
  any PCI and CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No